CLINICAL TRIAL: NCT02175927
Title: Prospective, Randomized Controlled Trial Comparing High Dose Amoxicillin Versus Tetracycline Based Quadruple Therapy as Second-line Treatment for Resistant Helicobacter Pylori Infection
Brief Title: High Dose Amoxicillin Versus Tetracycline as Second-line Treatment of Resistant Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Professor of GI Division, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2014007
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2015-12

CONDITIONS: Helicobacter Pylori Treatment Failure
Keywords: Helicobacter pylori; Treatment Failure; second-line therapy
MeSH Terms: interventions — Lansoprazole; Proton Pump Inhibitors; Bismuth; Metronidazole; Anti-Bacterial Agents; Amoxicillin; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Amoxicillin (Experimental): High dose amoxicillin/metronidazole-based quadruple therapy for 14 days: Lansoprazole 30mg bid, Bismuth Potassium Citrate 220mg bid, Amoxicillin 1000mg tid, Metronidazole 400mg qid
  Interventions: Drug: Lansoprazole; Drug: Bismuth Potassium Citrate; Drug: Metronidazole; Drug: Amoxicillin
- Tetracycline (Active Comparator): Classical quadruple therapy for 14 days: Lansoprazole 30mg bid, Bismuth Potassium Citrate 220mg bid, Tetracycline 500mg qid, Metronidazole 400mg qid
  Interventions: Drug: Lansoprazole; Drug: Bismuth Potassium Citrate; Drug: Metronidazole; Drug: Tetracycline

INTERVENTIONS:
Drug: Lansoprazole — antisecretory drug of each quadruple therapy
  Other Names: proton pump inhibitor
Drug: Bismuth Potassium Citrate — one component of each quadruple therapy
  Other Names: Bismuth
Drug: Metronidazole — antibiotic of each quadruple therapy
  Other Names: antibiotic
Drug: Amoxicillin — antibiotic of high dose amoxicillin based quadruple therapy
  Other Names: antibiotic
  Arms: High Dose Amoxicillin
Drug: Tetracycline — antibiotic of classical quadruple therapy
  Other Names: antibiotic
  Arms: Tetracycline

SUMMARY:
No trial has examined the the efficacy of high dose amoxicillin based quadruple therapy as second-line treatment for Helicobacter pylori infection. The study aims to compare the effectiveness and safety of 14-day high dose amoxicillin-based quadruple regiment with classical quadruple regiment for rescue eradication of Helicobacter pylori.

DETAILED DESCRIPTION:
Helicobacter pylori is the most successful human pathogen infecting an estimated 50% of the global population, and is associated with a spectrum of disease states, including chronic gastritis, duodenal and gastric ulcer, gastric adenocarcinoma, and gastric mucosa-associated lymphoid tissue lymphoma (MALToma).

Most Consensus Conferences and Clinical Guidelines recommend the prescription of a triple therapy including a proton pump inhibitor (PPI) and clarithromycin with either amoxicillin or metronidazole, as first-line treatment. However, the effectiveness of these triple-therapy regimens seems to have diminished over time, largely as a result of emerging resistance of the organism to clarithromycin. Avoiding problems due to antibiotic resistance has become an important issue when deciding a second-line rescue therapy for H. pylori infection

Bismuth-containing quadruple therapies have been used widely in second-line therapy of H. pylori infection, and are recommended by the Maastricht IV Consensus Conference report. Quadruple therapy can achieve a high rate of eradication success as a second-line treatment. A meta-analysis of quadruple therapy showed that metronidazole resistance had limited effect on the outcome when adequate dosages and durations are used. This meta-analysis also showed that compliance with quadruple therapy is high. Classical bismuth-based quadruple therapy consists of a PPI, bismuth, tetracycline and metronidazole. This regiment meets the proposed criteria for a second-line treatment: it does not contain the key antibiotic of the original regimen (clarithromycin), the treatment is not affected by clarithromycin resistance, metronidazole resistance in vitro does not affect the outcome of quadruple therapy significantly, compliance with the regimen is high and the regimen is effective in most parts of the world. But this regiment has high rate of side effects because of tetracycline.

Amoxicillin has low resistance rate as well as low percentage of side effects. The replacement of tetracycline by high dose amoxicillin in classical bismuth-containing quadruple therapy may be a better choice. Therefore, we will do a randomized trial to compare the eradication rate of 14-day high dose amoxicillin and metronidazole based bismuth-containing quadruple therapy with classical quadruple therapy for second-line Helicobacter pylori treatment.

ELIGIBILITY:
Inclusion Criteria:

* all patients had failed H.pylori therapies including clarithromycin, metronidazole and/or amoxicillin (if not allergic) before
* indication of rescue H pylori eradication treatment
* Ability and willingness to participate in the study and to sign and give informed consent

Exclusion Criteria:

* patients less than 18 years old
* previous gastric surgery
* pregnancy or lactation
* major systemic diseases,
* administration of antibiotics, bismuth, antisecretory drugs in the preceding 8 weeks
* allergy to any one of the medication used in the quadruple regimens.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | 2 months
  Access eradication rate of H. pylori by intention to treat (ITT) and per-protocol (PP) analysis in each treatment group

SECONDARY OUTCOMES:
Frequency of side effects of each treatment | 2 months
  Score side effects as mild, moderate or severe according to their influence on daily activities

OTHER OUTCOMES:
Minimal inhibitory concentrations (MIC) of antibiotics against each helicobacter pylori clinical isolate | 2 months
  Determine MIC of amoxicillin, tetracycline, and metronidazole by the twofold agar dilution method.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Lu H, Zhang W, Graham DY. Bismuth-containing quadruple therapy for Helicobacter pylori: lessons from China. Eur J Gastroenterol Hepatol. 2013 Oct;25(10):1134-40. doi: 10.1097/MEG.0b013e3283633b57. PMID 23778309